CLINICAL TRIAL: NCT00886093
Title: A Phase 1, Open Label, Randomized, Single Dose, Cross-Over Study To Evaluate The Effect Of Food On PF-04447943 Pharmacokinetics In Healthy Adult Subjects
Brief Title: A Study To Evaluate Whether Food Affects The Plasma Drug Levels Of A 35 mg Single Dose Of PF-04447943 Taken Orally In Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: B0401006
Record Dates: First submitted 2009-04-21; First posted 2009-04-22 (Estimated); Last update posted 2009-07-02 (Estimated); Status verified 2009-06

CONDITIONS: Healthy
Keywords: pharmacokinetics, single dose, crossover, fed vs fasted state
MeSH Terms: interventions — 6-(4-methyl-1-(pyrimidin-2-ylmethyl)pyrrolidin-3-yl)-1-(tetrahydro-2H-pyran-4-yl)-1,5-dihydro-4H-pyrazolo(3,4-d)pyrimidin-4-one

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence 1 (Experimental)
  Interventions: Drug: PF-04447943
- Sequence 2 (Experimental)
  Interventions: Drug: PF-04447943

INTERVENTIONS:
Drug: PF-04447943 — 35 mg tablet of PF-04447943 taken in the fed state in Period 1 followed a week later by administration of the same tablet and dose taken in the fasted state in Period 2
  Arms: Sequence 1
Drug: PF-04447943 — 35 mg tablet of PF-04447943 taken in the fasted state in Period 1 followed a week later by administration of the same tablet and dose in the fed state in Period 2.
  Arms: Sequence 2

SUMMARY:
The purpose of the study is to compare the plasma drug levels of PF-04447943 when taken as a 35 mg tablet after a high fat meal compared to when taken after fasting. Healthy adult volunteers will receive a single dose of the drug once when fasted and again when fed. The safety and tolerability of the drug will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects, not of child bearing potential.
* Age 18-55 inclusive
* Total body weight >50 kg.

Exclusion Criteria:

* Evidence or history of clinical significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic diseases
* History of orthostatic blood pressure changes or orthostatic symptoms
* Greater than 7 drinks of alcohol per week for women and greater than 14 drinks per week for men
* Smoking more than 5 cigarettes per day

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2009-04; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic endpoints include plasma PF-04447943 area under the curve (AUC), maximum plasma concentration (Cmax) and time of maximum plasma concentration (Tmax). | Up to 96 hours after drug administration
Safety endpoints include vital signs, ECGs, clinical laboratory tests, clinical evaluations and examinations, and adverse events. | Up to 96 hours after drug administration

SECONDARY OUTCOMES:
No secondary outcomes | No secondary outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0401006&StudyName=A%20Study%20To%20Evaluate%20Whether%20Food%20Affects%20The%20Plasma%20Drug%20Levels%20Of%20A%2035%20mg%20Single%20Dose%20Of%20PF-04447943%20Taken%20Orally%20In%20Healthy%20Ad